CLINICAL TRIAL: NCT07328269
Title: Effects of Mulligan Mobilization in Comparison With Maitland Mobilization in Temporomandibular Joint Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/20
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Temporomandibular Joint Dysfunction
Keywords: Hypomobility; Mulligan Mobilization; Maitland Mobilization
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: Participant divided into Two groups Group A recieves Mulligan Mobilization and Group B receives Maitland Mobilization with baseline treatment of myofascial release of temporalis and masseter muscle and Rocabado's 6*6 exercise program.
Who Masked: Participant
Masking Description: Participant will just have an idea of two interventions not the one given to him/her.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Mobilization (Active Comparator): Experimental Group A-Mulligan Mobilization. Myofascial release of temporalis and masseter muscle, Rocabado 6*6 exercise program.
  Interventions: Procedure: Mulligan Mobilization
- Maitland Mobilization (Experimental): Experimental Group B-Maitland Mobilization. Myofascial release of temporalis and masseter muscle. Rocabado 6*6 exercise program.
  Interventions: Procedure: Maitland Mobilization

INTERVENTIONS:
Procedure: Mulligan Mobilization — Both Mulligan and Maitland mobilization techniques with Myofascial release of temporalis and masseter and Rocabado 6*6 exercise program are applied over a two-week period with six sessions in total, focusing on improving TMJ mobility and reducing pain.
  Group A Mulligan mobilization emphasizes active patient involvement combined with therapist-applied glides, including lateral, anterior, medial, and distraction glides performed for 5-10 seconds with 3-5 repetitions per session.
  These techniques enhance mouth opening, lateral deviation, protrusion, and joint space while reducing stiffness and pain. And baseline treatment of myofascial release of temporalis and masseter muscle and Rocabado's 6*6 exercise program
  Arms: Mulligan Mobilization
Procedure: Maitland Mobilization — Group B-Maitland mobilization relies on graded oscillatory movements (Grades I-III) for 5-10 seconds with 3-5 oscillations, targeting pain relief and mobility in the pain-free range. Lower grades (I-II) are used for acute pain with gentle oscillations, while higher grades (II-III) provide moderate mobilization to improve protrusion, lateral deviation, and joint capsule mobility.
  And baseline treatment of myofascial release of temporalis and masseter muscle and Rocabado's 6*6 exercise program.
  Arms: Maitland Mobilization

SUMMARY:
The temporomandibular joint dysfunction is the second most common musculoskeletal pain after back pain, causing jaw pain, restricted movement, and joint sounds. NPRS and millimeter ruler will be used for the assessment of patient. This study will compare the effects of Mulligan and Maitland mobilization, commonly used treatment, on pain and Temporomandibular joint mobility through a randomized controlled trial, involving 30 participants divided into two groups for treatment.

DETAILED DESCRIPTION:
The temporomandibular joint connects the mandible to the temporal bone near the ear's tragus and plays a key role in mastication. It involves joint or muscle pain, jaw movement limitation, and joint popping sound Risk factors include trauma, bruxism, arthritis, stress, and poor posture, while diagnosis is commonly made using the DC/TMD criteria, focusing on pain and intra-articular dysfunction. Manual therapy techniques widely used to restore joint function and reduce pain.

Among these, Mulligan's Mobilization combines therapist-applied glides with active patient movement, while Maitland mobilization uses graded oscillatory techniques to relieve pain and improve mobility.

This study aims to compare the effects of Mulligan and Maitland mobilization on pain reduction and TMJ hypomobility in adults with TMD.

A randomized controlled trial will be conducted over one year. 30 participants will be selected through purposive sampling and randomly divided into two groups.

The intervention will last two weeks, comprising 06 treatment sessions. Assessments will be conducted at baseline, after the third session, and at the end of the second week.

Treatment will include lateral, anterior, medial, and distraction glides, combined with Rocabado's 6x6 exercises to improve functional movement. Myofascial release for the temporalis and masseter muscles will also be applied.

ELIGIBILITY:
Inclusion criteria

* Age 19-44 years.
* Both Genders (Male and Female).
* Patients diagnosed with TMJ hypomobility using the Manual Functional Analysis questionnaire based on DC/TMD criteria.
* Individuals with myofascial pain, scoring above 5 on the NRS and pain upon palpation of at least two of eight masticatory and neck muscles.
* Subjects with acute TMD and myofascial pain unrelated to active inflammation, infection, or recent trauma for at least six months.

Exclusion criteria

* Hypermobility of TMJs.
* Pregnancy.
* History of rheumatic and inflammatory diseases.
* A history of temporomandibular disorders treatment within last three months.
* Acute trauma or injuries of face, head or cervical spine, neurological disorders, taking medication that could affect the musculoskeletal system.

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 2 weeks
  Pain will be measured through Numeric Pain Rating Scale. The scoring for NPRS involves a scale from 0 to 10, where 0 indicates no pain. The interpretation of scores is as follows: 0 to 3 for mild pain, 4 to 6 for moderate pain, and 7 to 10 for severe pain.
Temporomandibular joint Hypomobility | 2 weeks
  Mandibular movements were assessed using a millimeter ruler to measure depression (50-60 mm), protrusion (5 mm), and lateral deviation (12-15 mm). Any "click" sounds or deviations during movement were recorded. Jaw movements maintained upper and lower teeth contact.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Punjab Province, Pakistan